CLINICAL TRIAL: NCT01113775
Title: Right Ventricular Dysfunction in Acute Pulmonary Embolism as Assessed by Spiral CT Scan: Comparison With Transthoracic Echocardiography and Evaluation of Prognostic Value
Brief Title: Pulmonary Embolism: Multifunctional Assessment of Prognosis
Acronym: PE-MAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Collaborators: Clinical Research Unit (Ambiguous)
Responsible Party: Giancarlo Agnelli, University of Perugia
Other Study IDs: CRU Unipg 02-06
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2009-10

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; computed tomography
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- presence of right ventricle dysfunction
- absence of right ventricle dysfunction

SUMMARY:
This is a prospective, observational, multicenter study. The primary aim of the study is to assess the accuracy of spiral CT scan to detect right ventricular dysfunction as compared to current 'gold standard'in patients with pulmonary embolism. At the purpose of this study right ventricular dysfunction as assessed by transthoracic echocardiography and serum levels of troponin are considered as gold standard.

The secondary aim of the study is to assess the prognostic value of right ventricular dysfunction as assessed by spiral CT scan.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a common and life-threatening disease. The incidence of a first episode of PE in acute care hospitals in the United States has been found to be 0.23 per 1000 with in-hospital mortality ranging from 30%, in case of cardiogenic shock, to about 0% in absence of right ventricular overload or hemodinamic impairment (1). In the intermediate group of patients with right ventricular overload but no hemodinamic impairment, in hospital mortality has been assessed to be about 5%. Right ventricular dysfunction as assessed at echocardiography and serum levels of Troponin I and T have been proposed as qualifying criteria for the identification of a subgroup of patients with pulmonary embolism and no hemodinamic impairment at high risk for in-hospital death. These patients could potentially benefit from more aggressive treatment.

A number of studies reported in favor of the association between echocardiographic RVD and early adverse outcome (PE recurrence and mortality) in patients with acute PE (3-6). In-hospital mortality in PE patients with and without echocardiographic RVD has been found to be 18.4% and 5.7%, respectively, regardless of the hemodinamic status (3). In 126 patients with acute pulmonary embolism, Ribeiro et al. reported a 7.9% overall in-hospital mortality (7). Mortality was 14.3% in patients with severe RVD. In a cohort of 2454 unselected patients with acute pulmonary embolism included in the ICOPER registry, 2-week mortality was 15.9% in patients presenting with RVD in comparison to 8% in patients without RVD (8). In the MAPPET 10% of patients with RVD died within 30 days as compared to 4.1% of patients without (9). Recent data confirmed that patients with objectively confirmed PE, normal BP and echocardiographic evidence of RVD have a high incidence of adverse outcome and may potentially benefit from more aggressive treatment (10).

Troponin I and T levels have also been described to be associated with in-hospital mortality and adverse in-hospital outcome in patients with acute pulmonary embolism (13-15).

In small studies with helical CT, the ratio of the right ventricle to left ventricle short axis diameters (RV/LV) has been proposed as an accurate sign for the presence of RVD (16-19). In addition, other criteria have been proposed, including deviation of the interventricular septum and the ratio of the pulmonary artery to ascending aorta diameters. Also, the extent of PE (ie, thrombus burden in the pulmonary arteries) has been proposed as an important parameter for predicting RVD (20-21). In a recent retrospective study in 120 patients with pulmonary embolism, seven patients died of PE. Both the RV/LV ratio and the obstruction index were shown to be significant risk factors for 3-month mortality (p = 0.04 and 0.01, respectively). No such relationship was found for the ratio of the pulmonary artery to ascending aorta diameters (p= 0.66) or for the shape of the interventricular septum (p = 0.20). The positive predictive value for PE-related mortality with an RV/LV ratio greater than 1.0 was 10.1% (95% confidence interval [CI]: 2.9%, 17.4%). The negative predictive value for an uneventful outcome with an RV/LV ratio of 1.0 or less was 100% (95% CI: 94.3%, 100%). There was a 11.2-fold increased risk of dying of PE for patients with an obstruction index of 40% or higher (95% CI: 1.3, 93.6). The CT obstruction index (29% ± 17%) and the Miller index (43% ± 25%) were well correlated (r = 0.867, p < 0.0001) with an excellent concordance between investigators for both the CT index (r = 0.944, p < 0.0001) and the Miller index (r = 0.904, p < 0.0001). A CT obstruction index greater than 40% identified more than 90% of patients with right ventricular dilatation.

Aim of the study The primary aim of the study is to assess the accuracy of spiral CT scan to detect right ventricular dysfunction as compared to current 'gold standard'. At the purpose of this study right ventricular dysfunction as assessed by transthoracic echocardiography and serum levels of troponin are considered as gold standard.

The secondary aim of the study is to assess the prognostic value of right ventricular dysfunction as assessed by spiral CT scan.

Feasibility In order to reach 200 evaluable patients, the Radiology Units of the participating centers will be asked to alert local investigators regarding all the patients with CT scan positive for acute pulmonary embolism. Local investigators should take care of organizing transthoracic echocardiography and troponin levels.

Four centers are required in order to complete the study in one year.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with spiral CT scan positive for acute pulmonary embolism and with transthoracic echocardiography ± 6 hours from spiral CT scan and baseline troponin levels evaluation

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with spiral CT scan positive for acute pulmonary embolism and with transthoracic echocardiography ± 6 hours from spiral CT scan and baseline troponin levels evaluation.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Becattini, MD, Study Chair — University Of Perugia
Locations (1):
- Internal and Cardiovascular Medicine Department, Perugia, Italy